CLINICAL TRIAL: NCT05235958
Title: Vascular Effects of Non-linear Periodized Exercise Training in Sedentary Adults With Elevated Cardiovascular Risk - The VascuFit Project
Brief Title: VascuFit: Exercise and Vascular Aging
Acronym: VascuFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karsten Königstein (Other)
Collaborators: University of Basel (Other); QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor-Investigator, Karsten Königstein, Clinical Scientist, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VF_CTgov
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Endothelial Function; Aerobic Exercise; Middle-aged Adults Sedentary, Elevated CV-risk)
Keywords: endothelium; flow-mediated vasodilation; sedentary; cardiovascular risk; aerobic exercise; vascular ageing
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled training intervention (8-weeks) with assessment of changes in clinical and molecular vascular biomarkers compared to their baseline value before the intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training intervention (Experimental): 8 weeks of non-linear periodized aerobic exercise; 3 sessions per week; 1 hour per session; standardized warm-up; individual training intensity according to cardiorespiratory fitness level
  Interventions: Other: non-linear periodized exercise (NLPE)
- Control Intervention (Sham Comparator): Recommendation to continue with current lifestyle (especially physical activity habits) during the following 8 weeks. At the final assessment after 8 weeks, individualized exercise recommendations according to established standard procedures in exercise medicine and offer to attend the standard medical follow-up in our outpatient clinics subsequent to study termination
  Interventions: Other: Exercise counselling

INTERVENTIONS:
Other: non-linear periodized exercise (NLPE) — Aerobic training derived from professional sports, that is characterized by variable periodization of training frequency, volume and intensity according to individual factors, such as physical and mental readiness, training progress and performance level
  Arms: Training intervention
Other: Exercise counselling — Standard recommendations for exercise and physical activity, that are individualized according to a medical health and fitness profile
  Arms: Control Intervention

SUMMARY:
Exercise is a cornerstone of health care helping to improve and maintain a good organ functionality, including vascular function, in health and disease. About twenty years ago, the introduction of high-intensity training has been a milestone in the evolution of exercise therapy by demonstrating the trainability of individuals independent of age and state of disease. Today, its practical implementation still faces barriers, such as lower physical and mental tolerance of exercise, long-term adherence and lack of individualization of training for optimal adaptations.

The proposed project is the logical next step to introduce non-linear periodized exercise training (NLPE), a method widely established in elite athletes, in exercise training of sedentary individuals. NLPE alternatingly involves person-centred periodization of training cycles and regeneration with high-intensity stimuli. It induces a broader range of physiological adaptations than moderate-intensity training while keeping a high compliance and without increasing the risk of overreaching. A study of patients with chronic-obstructive-pulmonary-disease and a study with resistance training of older adults indicated promising pulmonary and muscular effects. However, the effectiveness of NLPE to maintain and improve vascular function has not yet been assessed, although this may carry a huge clinical and socioeconomic potential by contributing to the reduction of cardiovascular morbidity and mortality.

VascuFit applies an 8-week training intervention to assess the effects of NLPE on the function of the vascular endothelium, measured by the non-invasive gold-standard method brachial arterial flow-mediated dilation (baFMD), in a sample of sedentary aging adults with cardiovascular risk factors. In addition, it will be the first study to measure training effects on a cluster of micro-ribonucleic acids (miRNAs) regulating key molecular pathways of endothelial (dys-)function. Thus, VascuFit aims to explore the potential of clinical and molecular biomarkers for the monitoring of individual vascular adaptability to a specific type of exercise. As a first step, this pilot-project is supposed to deliver proof-of-concept. Furthermore, it will generate important hypotheses to be addressed by exercise physiologists, medical professionals and biologists concerned with the optimization of individual training adaptations as well as utility and implementation of targeted training approaches in the health care of aging adults.

VascuFit aims to demonstrate the potential of NLPE as a training regimen to improve vascular function in sedentary individuals with elevated cardiovascular risk. This project may be the initial spark to raise exercise training to the next level, which is clearly necessary to sustainably strengthen the vascular capacities of "young" aging individuals.

DETAILED DESCRIPTION:
A detailed description of the study can be found at:

DOI: 10.1186/s12872-022-02905-1

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent, documented by signature
2. sedentary lifestyle, as not performing exercise on a regular basis and reaching less than the recommended 7.5 MET hours of at least moderate intensity activity per week
3. being mentally and physically able to attend and keep up training during the whole intervention period.

Exclusion Criteria:

1. current or chronic condition limiting exhaustive exercise (e.g. heart failure, infection, pulmonary disease)
2. any condition with elevated risk of a serious adverse event during exhaustive exercise (e.g. cardiomyopathy, acute myocardial infarction, stroke, uncontrolled hypertensive resting blood pressure ≥160/100mmHg)
3. chronic condition with severe affection of the vascular system (e.g. severe atherosclerosis, severe chronic kidney disease, autoimmune vasculitis, insulin dependent diabetes mellitus)
4. inability to follow advice during measurements and training sessions (e.g. language barriers, psychological disorders, dementia)
5. previous enrollment into the current study or participation in another study in the last four weeks.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Brachial-arterial flow-mediated vasodilation (baFMD) | 8 weeks
  Non-invasive ultrasound-based measurement of endothelial responsiveness of the brachial artery to an hyperemic stimulus. Changes of baFMD after the 8-week study period in comparison to the pre-intervention baseline values will be assessed.

SECONDARY OUTCOMES:
endomiR | 8 weeks
  Quantification of several micro-RNAs involved in key-regulatory pathways of the endothelial function of the macrovascular circulation. Changes of this micro-RNA cluster (endomiR) after the 8-week study period in comparison to the pre-intervention baseline values will be assessed.

OTHER OUTCOMES:
Static retinal vessel analysis (SVA) | 8 weeks
  Non-invasive ultrasound-based measurement of endothelial responsiveness of the retinal arterioles and venules. Changes of SVA after the 8-week study period in comparison to the pre-intervention baseline values will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Königstein, Dr. med., Principal Investigator — University of Basel
Locations (1):
- Departement of Sport, Exercise and Health, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After publication of the results, anonymized data and analytic codes may be shared upon request by the principal investigator (Dr. K. Königstein)
Supporting Information: Analytic Code
Time Frame: After publication of the study results.
Access Criteria: Justified request to the principle investigator (Dr. K. Königstein), i.e. reproduction of the study results, meta-analysis about a related scientific problem/question., data sampling for a big data project.

REFERENCES:
- [Derived] Konigstein K, Meier J, Angst T, Maurer DJ, Kropfl JM, Carrard J, Infanger D, Baumann S, Bischofsberger I, Harder M, Jaggi Y, Wettach S, Hanssen H, Schmidt-Trucksass A. VascuFit: vascular effects of non-linear periodized exercise training in sedentary adults with elevated cardiovascular risk - protocol for a randomized controlled trial. BMC Cardiovasc Disord. 2022 Oct 27;22(1):449. doi: 10.1186/s12872-022-02905-1. PMID 36303113